CLINICAL TRIAL: NCT01022112
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Dose-Ranging Study in Subjects With Type 2 Diabetes Mellitus to Evaluate the Efficacy, Safety, and Tolerability of Orally-Administered SGLT2 Inhibitor TA-7284
Brief Title: An Efficacy, Safety, and Tolerability Study for TA-7284 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-7284-04
Record Dates: First submitted 2009-11-29; First posted 2009-12-01 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: TA-7284; JNJ-28431754; Canagliflozin; Type 2 diabetes mellitus; Sodium Glucose Co-transporter (SGLT2 inhibitor)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- TA-7284-Low (Experimental)
  Interventions: Drug: TA-7284-Low
- TA-7284-Low-middle (Experimental)
  Interventions: Drug: TA-7284-Low-middle
- TA-7284-High-middle (Experimental)
  Interventions: Drug: TA-7284-High-middle
- TA-7284-High (Experimental)
  Interventions: Drug: TA-7284-High
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TA-7284-Low — TA-7284-Low
  Arms: TA-7284-Low
Drug: TA-7284-Low-middle — TA-7284-Low-middle
  Arms: TA-7284-Low-middle
Drug: TA-7284-High-middle — TA-7284-High-middle
  Arms: TA-7284-High-middle
Drug: TA-7284-High — TA-7284-High
  Arms: TA-7284-High
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy, safety, and tolerability of TA-7284 compared with placebo in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is well recognized as a major public health problem that presents patients with a significant risk of complications including heart disease, retinopathy, nephropathy, and neuropathy. Various classes of orally administered antihyperglycemic agents have been developed for the treatment of T2DM and although individual agents may be highly effective for some patients, it is still difficult to maintain optimal glycemic control in most patients, resulting in high rates of morbidity and mortality in the diabetic population. This is a randomized, double-blind, placebo-controlled, parallel-group study to demonstrate the efficacy, safety, and tolerability of TA-7284 compared with placebo in patients with T2DM, who are not optimally controlled on diet and exercise. The primary study hypothesis is that the study drug will be superior to placebo as assessed by the change in HbA1c from baseline. The patients will receive tablets of TA-7284, or placebo, once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 20 to 80 years inclusive on the day of informed consent;
* Patients who was diagnosed with type 2 diabetes mellitus at least 3 months before the start of the run-in period;
* Patients with HbA1c of ≥6.5% and ≤9.5% (according to the Japan Diabetic Society [JDS] criteria) on the start day of the run-in period;

Exclusion Criteria:

* Type I diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes mellitus (acromegaly, Cushing's syndrome, etc.);
* Past or current history of severe diabetic complications (proliferative diabetic retinopathy, stage III or later stage overt nephropathy, diabetic ketoacidosis, or serious diabetic neuropathy);
* Fasting blood glucose of >270 mg/dL on the start day of the run-in period or at Week 2 of the run-in period;
* eGFR of <60 mL/min/1.73 m2 on the start day of the run-in period;
* Systolic blood pressure of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg on the start or end day of the run-in period;
* History of myocardial infarction, unstable angina, or cerebrovascular disorder within 3 months before the start of the run-in period;
* Concurrent serious (e.g., requiring inpatient hospitalization or surgical intervention) renal or hepatic disease;
* Past or current history of malignant tumor; however, this criterion shall not apply to those who have been free of relapse for at least 5 years even with a history of malignant tumor.
* Past or current history of drug hypersensitivity such as shock and anaphylactoid symptoms;
* Pregnant women, lactating mothers, or women of childbearing potential;
* Any condition that subjects are assessed to be ineligible by the investigator (sub investigator).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuya Inagaki, M.D., Study Director — Kyoto University, Graduate School of Medicine; Kazuoki Kondo, M.D., Study Director — Tanabe Pharma Corporation; Tadashi Yoshida, M.D., Study Director — Tanabe Pharma Corporation
Locations (6):
- Japan (6):
  - Research site, Chugoku
  - Research site, Kanto
  - Research site, Kinki
  - Research site, Kyushu
  - Research site, Shikoku
  - Research site, Tōhoku

RESULTS

PARTICIPANT FLOW:
Groups:
- TA-7284-Low: TA-7284 50 mg, once daily for 12 weeks
- TA-7284-Low-middle: TA-7284 100 mg, once daily for 12 weeks
- TA-7284-High-middle: TA-7284 200 mg, once daily for 12 weeks
- TA-7284-High: TA-7284 300 mg, once daily for 12 weeks
- Placebo: TA-7284 Placebo, once daily for 12 weeks
Period: Overall Study
Arm/Group | TA-7284-Low | TA-7284-Low-middle | TA-7284-High-middle | TA-7284-High | Placebo
Started | 82 | 74 | 77 | 75 | 75
Completed | 79 | 71 | 74 | 72 | 65
Not Completed | 3 | 3 | 3 | 3 | 10
Not completed — Adverse Event | 1 | 2 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2 | 1
Not completed — Fasting plasma glucose level increased | 1 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TA-7284-Low | TA-7284-Low-middle | TA-7284-High-middle | TA-7284-High | Placebo | Total
Number analyzed (Participants) | 82 | 74 | 77 | 75 | 75 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.8) | 57.7 (10.5) | 57 (10.6) | 57.1 (10.1) | 57.7 (11.0) | 57.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 22 | 27 | 20 | 21 | 122
  Male | 50 | 52 | 50 | 55 | 54 | 261

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (A1C) From Baseline (NGSP Value)
Time Frame: 12 weeks
Population: Full analysis set, last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percent HbA1C
Arm/Group | TA-7284-Low | TA-7284-Low-middle | TA-7284-High-middle | TA-7284-High | Placebo
Number analyzed (Participants) | 82 | 74 | 75 | 75 | 75
percent HbA1C | -0.61 (0.06) | -0.80 (0.06) | -0.79 (0.06) | -0.88 (0.06) | 0.11 (0.06)

2. Secondary Outcome: Fasting Blood Glucose, Body Weight
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Safety and Tolerability
Time Frame: 14 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | TA-7284-Low | TA-7284-Low-middle | TA-7284-High-middle | TA-7284-High | Placebo
Serious Adverse Events (participants affected / at risk) | 1/82 | 0/74 | 0/77 | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 36/82 | 34/74 | 38/77 | 34/75 | 26/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-7284-Low (N=82) | TA-7284-Low-middle (N=74) | TA-7284-High-middle (N=77) | TA-7284-High (N=75) | Placebo (N=75)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-7284-Low (N=82) | TA-7284-Low-middle (N=74) | TA-7284-High-middle (N=77) | TA-7284-High (N=75) | Placebo (N=75)
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 8 | 10 | 8 | 9 | 10
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Stitch abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 1 | 0
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 1 | 1 | 3 | 2 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 2 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 3 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vulvar erosion (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2
Hunger (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 3 | 0 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 1 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood ketone body increased (Investigations) | 4 | 5 | 9 | 6 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 2 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 0 | 0
Urine output increased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other